CLINICAL TRIAL: NCT01516606
Title: Phase II Clinical Trial on the Activity of Salvage Therapy With High Dose Oral Clarithromycin in Patients With Relapsed or Refractory Extranodal Marginal Zone Lymphoma
Brief Title: Salvage Therapy With High Dose Oral Clarithromycin in Relapsed or Refractory Extranodal Marginal Zone Lymphoma
Acronym: HD-K
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andres J. M. Ferreri (Other)
Responsible Party: Sponsor-Investigator, Andres J. M. Ferreri, MD, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HD-K
Record Dates: First submitted 2012-01-06; First posted 2012-01-25 (Estimated); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Lymphoma
Keywords: MALT; refractory; relapsed; extranodal; relapsed or refractory extranodal marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Recurrence | interventions — Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- clarithromycin, oral, high dose (Experimental): 2 g/day clarithromycin (once a day) for 14 days followed by 7 days interval to be repeated for 4 cycles in total
  Interventions: Drug: clarithromycin, oral, high dose

INTERVENTIONS:
Drug: clarithromycin, oral, high dose — 2 g/day clarithromycin (once a day) for 14 days followed by 7 days interval to be repeated for 4 cycles in total
  Other Names: klacid

SUMMARY:
This is a prospective, phase II study on the activity and tolerability of high dose (2 g/day) oral clarithromycin for the treatment of relapsed or refractory extranodal marginal zone lymphoma.

DETAILED DESCRIPTION:
A 6-month regimen of oral clarithromycin has been associated with a 35% ORR in patients with relapsed/refractory marginal zone B-cell lymphoma. Responses were more common among patients with conjunctival lymphoma. This could be explained at least in part by the elimination of clarithromycin by tears, suggesting that a higher tumor bioavailability of this antibiotic could result in a higher activity. Thus, a higher dose of clarithromycin could be associated with a higher tumor bioavailability in tissues other than the conjunctiva.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed diagnosis of extranodal extra-gastric marginal zone cell B lymphoma or gastric Helicobacter pylori positive lymphoma refractory to conventional antibiotic therapy, or H. pylori negative
* at least one measurable lesion
* relapsed or refractory lymphoma after systemic (chemotherapy, immunotherapy, antibiotic) or local (surgery or radiation) therapy
* ECOG PS </= 3
* no prior antibiotic therapy within 3 months before enrollment

Exclusion Criteria:

* HIV 1-2 infection
* concomitant conventional or experimental antitumor therapy (chemotherapy, radiotherapy, immunotherapy, corticosteroids)
* severe inadequate liver (AST </=3 ULN, ALT </= 3 ULN, bilirubin </=3 ULN) or renal (creatinine </= 1.5 ULN) function
* allergy to macrolides
* concomitant malignant neoplasms within prior 5 years (with the exclusion of basal cell carcinoma, in situ spinocellular carcinoma of skin and cervix)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
assessment of responses | The best clinical response at 6 months from trial registration
  evaluation of activity in terms of global responses, complete responses and duration of responses

CONTACTS AND LOCATIONS:
Overall Officials: Andrés JM Ferreri, MD, Study Chair — San Raffaele Scientific Institute, Milano, Italy
Locations (1):
- Dpt of OncoHematology - Fondazione Centro San Raffaele del Monte Tabor, Milan, Italy

REFERENCES:
- [Derived] Ferreri AJ, Sassone M, Kiesewetter B, Govi S, Scarfo L, Donadoni G, Raderer M. High-dose clarithromycin is an active monotherapy for patients with relapsed/refractory extranodal marginal zone lymphoma of mucosa-associated lymphoid tissue (MALT): the HD-K phase II trial. Ann Oncol. 2015 Aug;26(8):1760-5. doi: 10.1093/annonc/mdv214. Epub 2015 May 1. PMID 25935794